CLINICAL TRIAL: NCT07349511
Title: Diagnostic Validity of a Quantitative Pulp Pain Scoring System and Its Association With Postoperative Clinical Outcomes: A Prospective Study
Brief Title: Diagnostic Validity of a Quantitative Pulp Pain Scoring System and Its Association With Postoperative Clinical Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Medine Ciçek, endodontist, Recep Tayyip Erdogan University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MÇ
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain After Endodontic Treatment; Direct Pulp Capping; Vital Pulp Therapy
Keywords: pulpitis; postoperative pain; vital pulp therapy; pulp capping; root canal treatment
MeSH Terms: conditions — Pulpitis; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: a prospective clinical study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vital pulp therapy (Experimental): In this study, treatment planning was based on the total score obtained from the Youden symptom scoring system. Patients with scores below 25 were diagnosed with reversible pulpitis and treated with vital pulp therapy. Indirect pulp capping was performed in cases where no pulp exposure occurred during caries removal. Direct pulp capping was performed in cases where pulp exposure occurred during caries removal but the clinical and symptomatic findings were consistent with a diagnosis of reversible pulpitis.
  Interventions: Other: Vital pulp therapy procedure based on the total score obtained from the Youden symptom scoring system
- root canal treatment (Experimental): Patients with scores of 25 or higher were diagnosed with irreversible pulpitis and treated with root canal therapy, to ensure standardized and reproducible treatment allocation.
  Interventions: Other: Root canal treatment procedure based on the total score obtained from the Youden symptom scoring system

INTERVENTIONS:
Other: Root canal treatment procedure based on the total score obtained from the Youden symptom scoring system — All procedures were performed under rubber dam isolation, in a single visit, and by a single operator. For root canal treatment, pulp extirpation was performed after access cavity preparation and canals were shaped with rotary nickel-titanium instruments. A standardized irrigation protocol was applied using 2.5% sodium hypochlorite during and after instrumentation, followed by 17% EDTA for smear layer removal. All irrigants were activated by passive ultrasonic irrigation in three 20-second cycles. After irrigation, canals were dried with sterile paper points and obturated with gutta-percha and a resin-based sealer using the cold lateral compaction technique. All teeth received permanent coronal restorations.
  Arms: root canal treatment
Other: Vital pulp therapy procedure based on the total score obtained from the Youden symptom scoring system — All procedures were performed under rubber dam isolation, in a single visit, and by a single operator. Indirect pulp capping was performed in cases where no pulp exposure occurred during caries removal. In teeth with deep dentin caries but preserved pulpal integrity, all carious tissue was removed while maintaining a thin layer of dentin adjacent to the pulp, and indirect pulp capping was subsequently performed. After confirming the absence of pulp exposure through clinical examination, mineral trioxide aggregate (MTA) was applied to the dentin surface adjacent to the pulp.
  Direct pulp capping was performed in cases where pulp exposure occurred during caries removal but the clinical and symptomatic findings were consistent with a diagnosis of reversible pulpitis. Following pulp exposure, hemostasis was achieved. After adequate hemostasis was obtained, MTA was applied to the exposed pulp tissue. Permanent coronal restoration of all teeth were performed.
  Arms: vital pulp therapy

SUMMARY:
Pulpal diseases are among the most common reasons for endodontic treatment in dental practice. The dental pulp plays a critical role in maintaining tooth vitality, and its pathological changes directly affect pain perception and patient quality of life. Therefore, accurate diagnosis of pulpal diseases is essential for patient-centered treatment planning. Distinguishing between reversible and irreversible pulpitis remains a major diagnostic challenge in endodontics, as this distinction relies largely on subjective symptom characteristics that vary considerably among patients. This uncertainty particularly affects newly graduated dentists, highlighting the need for objective and reproducible diagnostic tools in both dental education and clinical practice.

To address these challenges, several classification systems for pulpal disease assessment have been proposed. Recently, Kumar et al. introduced the Pulp Pain Assessment Tool, a validated 11-item scoring system that quantifies both the intensity and qualitative aspects of pulpal pain. This tool generates scores ranging from 11 to 44, with a statistically determined cut-off value of 25 to differentiate reversible from irreversible pulpitis, providing a reproducible and standardized diagnostic framework.

Although this quantitative approach may improve diagnostic objectivity and clinical decision-making, its agreement with established systems such as the American Association of Endodontists (AAE) classification and the Wolters diagnostic framework has not yet been systematically evaluated. Therefore, the primary aim of this study was to assess the diagnostic validity of Kumar's pulp pain assessment tool and its concordance with the AAE and Wolters classification systems. The secondary aim was to evaluate the relationship between total symptom scores and postoperative outcomes, including pain levels and analgesic consumption, according to the type of treatment performed (vital pulp therapy or root canal treatment).

The null hypotheses were that there would be no significant difference in diagnostic agreement among the AAE classification, the Wolters system, and Kumar's scoring model, and that total symptom scores would not be associated with postoperative pain or analgesic consumption.

DETAILED DESCRIPTION:
Material and methods This prospective, single-center observational clinical study aimed to evaluate the diagnostic concordance of a quantitative symptom-based scoring system for pulpal symptom severity and its association with patient-centered clinical outcomes. Ethical approval was obtained from the Recep Tayyip Erdoğan University Non-Interventional Clinical Research Ethics Committee (2025/435), and written informed consent was obtained from all participants.

The study was conducted at the Department of Endodontics, Faculty of Dentistry, Recep Tayyip Erdoğan University. All consecutive patients presenting with acute dental complaints were screened, and those meeting the predefined inclusion criteria were enrolled following clinical and radiographic examinations.

Patient selection Eligible participants were adults (≥18 years) presenting with acute symptoms related to a single vital tooth without clinical or radiographic evidence of periapical pathology. Exclusion criteria included pulpal necrosis, previously root canal-treated teeth, non-pulpal periapical pathology, regular use of analgesic or anti-inflammatory drugs, pregnancy, immunosuppressive conditions, and systemic diseases affecting pain perception, healing, or follow-up.

Classification of Pulpal Diseases and Diagnostic Criteria Pulpal status was independently evaluated at the time of presentation using three diagnostic approaches.

Wolters Diagnostic Classification Pulpal inflammation was classified according to the four-level system proposed by Wolters et al. as initial, mild, moderate, or severe pulpitis, based on the biological continuity and severity of symptoms [4]. Initial and mild pulpitis-characterized by reversible, stimulus-related pain without significant spontaneous symptoms-were categorized as reversible pulpitis, whereas moderate and severe pulpitis-defined by intense, prolonged, and often spontaneous pain affecting daily activities-were categorized as irreversible pulpitis. This classification was based on clinical parameters including response duration to thermal stimuli, spontaneous pain, analgesic requirement, and impact on daily life.

AAE Diagnostic Classification Pulpal diagnosis was also performed according to the American Association of Endodontists (AAE) classification [2], based on patient history, thermal and electric pulp testing, and the presence of spontaneous pain. Pulpal conditions were categorized as normal pulp, reversible pulpitis, irreversible pulpitis (symptomatic or asymptomatic), or pulpal necrosis, with diagnostic decisions relying on clinical findings and symptom interpretation.

Kumar et al.'s Pulp Pain Assessment Tool (PPAT) In this study, the validated Pulp Pain Assessment Tool developed by Kumar et al. was used to quantitatively assess pulpal symptom severity [3]. The tool consists of 11 items and generates a total score ranging from 11 to 44. A cutoff value of 25-established through receiver operating characteristic analysis and the Youden index in the original validation study-was used to differentiate reversible from irreversible pulpitis.

The first five items assess pain intensity using the Numeric Rating Scale-11 (NRS-11) under different conditions (rest, cold, heat, sweet stimuli, and lying down). NRS-11 scores were categorized as no pain (0), mild (1-3), moderate (4-6), or severe (7-10) and converted into numerical scores ranging from 1 to 4.

The remaining six items evaluate pain characteristics, including spontaneity, duration, radiation, positional changes, pain on biting, and analgesic requirement, using a four-point Likert scale (1 = never to 4 = most of the time/continuously). Scores from all items were summed to obtain a total symptom score, which was considered a quantitative indicator of overall pulpal symptom severity.

Treatment Algorithm and Clinical Protocols Treatment allocation was standardized according to the total score obtained from the Youden symptom-based scoring system. Patients with scores <25 were diagnosed with reversible pulpitis and treated with vital pulp therapy, whereas those with scores ≥25 were diagnosed with irreversible pulpitis and treated with root canal therapy. All procedures were performed under rubber dam isolation, in a single visit, and by a single operator to minimize operator-related variability.

Indirect Pulp Capping Indirect pulp capping was performed in teeth without pulp exposure during caries removal. After complete caries excavation while preserving a thin dentin layer adjacent to the pulp, mineral trioxide aggregate (MTA) (Angelus Bio-C Repair, Londrina, Brazil) was applied to the affected dentin.

Direct Pulp Capping Direct pulp capping was carried out in cases of pulp exposure consistent with a diagnosis of reversible pulpitis. The number, size, and location of exposure sites were recorded. Hemostasis was achieved and bleeding control time was documented before application of MTA (Angelus Bio-C Repair, Londrina, Brazil) to the exposed pulp tissue.

Root Canal Treatment For teeth undergoing root canal treatment, pulp extirpation was performed using #10-15 K-type hand files following access cavity preparation. Working length was determined using an electronic apex locator (Woodpex 5, Woodpecker, China), and canals were shaped with rotary nickel-titanium instruments (EndoArt Smart Gold, İnci Dental, Turkey) operated at 300 rpm and 2-5.2 Ncm torque using a torque-controlled motor.

Following canal shaping, a standardized irrigation protocol was applied. Each canal was irrigated with 2.5% sodium hypochlorite during and after instrumentation (total volume: 10 mL per canal), followed by 17% EDTA (2 mL for 1 minute) to remove the smear layer. All irrigating solutions were activated using passive ultrasonic irrigation in three 20-second cycles.

After irrigation, canals were dried with sterile paper points and obturated using a resin-based sealer and gutta-percha cones with the cold lateral compaction technique. All teeth treated with vital pulp therapy or root canal treatment received permanent coronal restorations using a self-etch adhesive system and composite resin, ensuring adequate coronal sealing.

Cases with iatrogenic complications, such as perforation or instrument separation, were excluded. Clinical parameters, including pulp exposure characteristics, bleeding duration, and total treatment time, were systematically recorded using standardized data collection forms.

Postoperative Pain and Analgesic Follow-up Postoperative pain intensity was assessed using the Visual Analog Scale (VAS), and a VAS score greater than 0 was considered indicative of the presence of postoperative pain. Following treatment, the use of the VAS scale was explained to all patients in detail, and both written and verbal instructions were provided regarding how pain assessment should be performed at each designated time interval.

Within the follow-up protocol, patients were not asked to record a single point-in-time pain score at the specified time points. Instead, they were instructed to record the maximum pain intensity experienced within each predefined time interval. Accordingly, patients were asked to document the highest level of pain they experienced using the VAS scale during the following postoperative time intervals: 0-8 hours, 8-24 hours, 24-48 hours, 48-72 hours, 72-120 hours, and 120-168 hours after treatment. In cases where patients felt the need to take an analgesic during any of these intervals, they were specifically instructed to record the maximum pain intensity experienced immediately prior to analgesic intake on the VAS form.

Postoperative analgesic use was recorded on a per-patient basis as yes or no. Patients who used analgesics were additionally instructed to document the timing of use, the type of medication taken, and the frequency of intake. All patients were prescribed paracetamol as the first-line analgesic for postoperative pain management.

Patients were scheduled for a clinical follow-up visit 7 days after treatment. In addition, to minimize patient attrition and data loss during the follow-up period, patients were contacted by telephone at time points close to the scheduled assessment intervals. During these communications, patients were reminded to complete their VAS forms, and information regarding analgesic use was verified. This follow-up strategy was implemented to enhance patient compliance during the postoperative period and to achieve the highest possible level of data completeness within the study.

Interobserver reliability At the time of clinical presentation, patients were independently assessed for pulpal status by two different observers using the Youden symptom scoring system. One observer was a fifth-year dental student at the graduation stage, and the other was an endodontic specialist with six years of clinical experience. Both observers recorded the clinical and symptomatic findings of the patients according to the diagnostic systems defined in the study, without being aware of each other's evaluations.

Because the majority of patients presented with acute dental complaints and immediate initiation of treatment following diagnosis was clinically mandatory, it was not feasible to allow the required time interval for an intraobserver (test-retest) reliability assessment, which would have required re-evaluation after approximately four weeks. Therefore, only interobserver reliability analysis was performed in this study.

Interobserver diagnostic agreement was evaluated based on the binary diagnostic categories (reversible versus irreversible pulpitis) derived from the Youden score. Agreement between observers was calculated using Cohen's kappa coefficient, which is appropriate for categorical data. Kappa values were reported together with their 95% confidence intervals. In addition, the McNemar test was applied to assess potential systematic differences in diagnostic distributions between the two observers.

Statistical Analysis All statistical analyses were performed using Python (version 3.14), primarily with the pandas, numpy, and statsmodels libraries. Continuous variables were summarized using mean ± standard deviation and median (interquartile range), while categorical variables were presented as frequencies and percentages. The Kumar et al.'s Pulp Pain Assessment Tool was treated as a continuous variable and its distribution was descriptively examined across different clinical classification systems to illustrate how symptom severity mapped onto the scoring continuum. Agreement between diagnostic classification systems was evaluated using percent agreement and Cohen's kappa statistics, and asymmetry in discordant classifications was assessed using McNemar's test.

Postoperative pain intensity was assessed longitudinally using VAS scores measured at multiple postoperative time points. For each treatment group, the proportion of patients reporting pain (VAS > 0) and the proportion using analgesics were calculated at each time point and visualized to describe temporal trends. To identify factors associated with pain severity while accounting for repeated measurements within individuals, generalized estimating equation (GEE) models with a Gaussian family and robust standard errors were applied separately for VPTand RCT(RCT) groups. Time was modelled as a categorical variable with the earliest postoperative assessment as the reference. An autoregressive working correlation structure was used, with alternative structures considered when necessary to ensure model stability. In addition, for VPT cases, multivariable logistic regression models were constructed to explore factors associated with binary outcomes (presence of postoperative pain and analgesic use). To minimize model instability, variables with sparse categories were excluded when appropriate, and missing values in continuous procedure-related variables were handled using median imputation. A two-sided p value < 0.05 was considered statistically significant for all analyses.

ELIGIBILITY:
Inclusion Criteria: Patients aged 18 years or older presenting with acute symptoms associated with a single tooth exhibiting vital pulp tissue, without clinical or radiographic evidence of periapical pathology, and who consented to participate were included.

Exclusion Criteria: Exclusion criteria comprised pulpal necrosis, previously root canal-treated teeth, periapical pathology unrelated to pulpal disease, regular use of analgesic or anti-inflammatory medications, pregnancy, immunosuppressive conditions, and systemic diseases that could interfere with pain perception, healing, or follow-up compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2025-11-04 (Actual); Primary Completion 2026-01-01 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
Diagnostic concordance of the Pulp Pain Assessment Tool (PPAT) with established pulpal diagnostic systems | At baseline (at the time of patient presentation, prior to treatment)
  Diagnostic agreement between the Pulp Pain Assessment Tool (PPAT) and the American Association of Endodontists (AAE) classification and the Wolters diagnostic system for pulpal disease, evaluated using Cohen's kappa coefficient.

SECONDARY OUTCOMES:
Postoperative pain intensity | Up to 7 days after treatment
  Postoperative pain intensity assessed using the Visual Analog Scale (VAS). Patients recorded the maximum pain intensity experienced during predefined postoperative intervals (0-8 h, 8-24 h, 24-48 h, 48-72 h, 72-120 h, and 120-168 h) following treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdoğan University Faculty of Dentistry, Department of Endodontics, Rize, Centre, Turkey (Türkiye)